CLINICAL TRIAL: NCT07284446
Title: Prevalence of Depressive Symptoms and Cognitive Impairment and Their Association With Worse Outcomes in a Cohort of Hospitalized Patients With Chronic Heart Failure
Brief Title: Depressive Symptoms, Cognitive Impairment, and Outcomes in Hospitalized Chronic Heart Failure Patients
Acronym: DSCI-CHF
Status: Recruiting | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Andrius Ališauskas, MD, Principal Investigator, Lithuanian University of Health Sciences
Other Study IDs: PEACE-pro-HF-1
Record Dates: First submitted 2025-11-22; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Congestive Heart Failure Chronic; Cognitive Impairment, Mild; Depressive Symptoms Mild to Moderate in Severity
Keywords: Congestive Heart Failure; Mild Cognitive Impairment; Long-term Outcomes; Mild Depressive Symptoms; Rehospitalizations
MeSH Terms: conditions — Cognitive Dysfunction; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CHF Group: Cohort of patients hospitalized due to Exacerbation of Chronic heart failure

SUMMARY:
The goal of this observational study is to learn about the prevalence of depressive symptoms and cognitive impairment and their association with worse outcomes in a cohort of hospitalized patients between the ages of 18 ang 85 years with chronic heart failure. The main question it aims to answer is:

• Does the presence of depressive symptoms and cognitive impairment lead to worse outcomes in a cohort of hospitalized patients with chronic heart failure? Participants who are hospitalized due to exacerbation of chronic heart failure will answer survey questions to assess their cognitive function and depressive symptoms.

DETAILED DESCRIPTION:
This is a single-centre, prospective, observational cohort study designed to evaluate the prevalence of depressive symptoms and cognitive impairment and to investigate their association with worse clinical outcomes in hospitalized patients with chronic heart failure (CHF). The study will be conducted at the Department of Cardiology and the Internal Medicine Department's Cardiology Profile of the Lithuanian University of Health Sciences Kaunas Hospital (LSMU Kaunas Hospital), Kaunas, Lithuania, where the majority of Kaunas region patients with CHF are admitted for inpatient care.

CHF is a common clinical syndrome resulting from structural and/or functional cardiac abnormalities, leading to typical symptoms, frequent hospitalizations, reduced quality of life, and high mortality. In addition to somatic burden, patients with CHF frequently experience cognitive impairment and mental health disorders, particularly anxiety and depressive disorders. These conditions are highly prevalent and are associated with poorer self-care, impaired adherence to therapy, diminished quality of life, and worse prognosis. Despite increasing recognition of their importance, depressive symptoms, anxiety, and cognitive impairment remain under-recognized and insufficiently integrated into routine CHF management. Symptom overlap between CHF and mental or cognitive disorders further complicates detection, contributing to underdiagnosis and undertreatment.

To address this gap, the present study will systematically assess depressive symptoms and cognitive function in a consecutively enrolled cohort of hospitalized patients with CHF and will examine how these factors relate to short- and medium-term outcomes.

The main objectives are:

1. to determine the prevalence of depressive symptoms in hospitalized patients with CHF;
2. to determine the prevalence of cognitive impairment in the same population;
3. to evaluate the association between depressive symptoms and worse CHF outcomes;
4. to evaluate the association between cognitive impairment and worse CHF outcomes.

The planned sample size is 300 patients, calculated on the basis of survival as the main clinical endpoint (mortality and CHF-related rehospitalizations), assuming an expected prevalence of depressive symptoms and cognitive impairment of approximately 10-20% among patients with CHF and a hazard ratio of 2.5 for adverse outcomes in patients with depressive symptoms and/or cognitive impairment compared with those without. Patient recruitment is anticipated to take approximately 24 months, with an additional 12 months of follow-up for clinical outcomes after the last patient is enrolled.

After clinical stabilization during the index hospitalization, eligible patients will provide written informed consent and a structured interview and baseline assessment will be performed approximately 48 hours after stabilization.

The assessment will include:

1. collection of demographic data;
2. physical examination;
3. anthropometric measurements;
4. completion of standardized, validated questionnaires for depressive symptoms and cognitive function.

Depressive symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9) and the Hospital Anxiety and Depression Scale (HADS), both in validated Lithuanian versions. Cognitive function will be assessed with the Lithuanian version of the Montreal Cognitive Assessment (MoCA). All questionnaires will be administered by the principal investigator or another physician-investigator working in the study centre. The same set of questionnaires (PHQ-9, HADS, MoCA) will be repeated on the last day of the hospital stay in order to evaluate the dynamics of depressive symptoms and cognitive function during hospitalization.

In addition, routine clinical, laboratory, and instrumental data will be extracted from the paper and electronic medical records. Information on in-hospital management, including pharmacological therapy and any procedures, will also be collected.

The primary clinical outcomes of interest are:

1. all-cause mortality during the index hospitalization;
2. all-cause mortality after discharge;
3. CHF-related rehospitalizations during the first 12 months after discharge from the index hospitalization.

The main exposures of interest are the presence and severity of depressive symptoms and cognitive impairment at baseline and at discharge, as defined by established cut-offs in PHQ-9, HADS, and MoCA scores.

Data will be recorded on paper case report forms and subsequently entered into a dedicated electronic database.

Statistical analyses will include descriptive statistics to characterize the prevalence and severity of depressive symptoms and cognitive impairment; univariable and multivariable regression models to examine associations between depressive symptoms and cognitive impairment and clinical and demographic characteristics; and survival analyses (Kaplan-Meier curves and Cox proportional hazards models) to evaluate the relationship between depressive symptoms, cognitive impairment, and time to death or CHF-related rehospitalization. A two-sided p value <0.05 will be considered statistically significant.

By quantifying the prevalence of depressive symptoms and cognitive impairment and clarifying their prognostic significance for patients hospitalized with CHF in Lithuania, this study aims to provide evidence to support more systematic screening, follow-up, and targeted psychosocial and cognitive interventions in this high-risk population. The findings may inform local and international clinical practice by highlighting the need to integrate mental health and cognitive assessment into comprehensive CHF management pathways.

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalized primarily for CHF exacerbation;
* clinically stable, able to provide informed consent;
* do not have severe cognitive impairment that would preclude valid questionnaire administration.

Exclusion Criteria:

* hospitalization for acute heart failure;
* total length of hospital stay <96 hours;
* absence of transthoracic echocardiography (TTE) within the last 12 months and no TTE planned;
* severe visual impairment preventing completion of the visual part of the Montreal Cognitive Assessment;
* refusal to participate.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized to the Department of Cardiology and the Internal Medicine Department's Cardiology Profile at the Lithuanian University of Health Sciences Kaunas Hospital, Kaunas, Lithuania
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2028-12-02 (Estimated); Study Completion 2028-12-02 (Estimated)

PRIMARY OUTCOMES:
In-hospital all-cause mortality | From enrollment to the end of treatment up to 30 days
  Lethal all-cause outcome
In-hospital MACE | From enrollment to the end of treatment up to 30 days
  In-hospital Major Adverse Cardiovascular Event (including myocardial infarction, stroke, cardiovascular death, and need for revascularization [like repeat PCI or bypass surgery])
Number of Participants with chronic heart failure-related rehospitalization | 12 months post discharge from the hospital
  Subsequent hospitalization due to chronic heart failure exacerbation (decompensation) within 12 months after the index admission to the hospital (enrollment to the study)

CONTACTS AND LOCATIONS:
Overall Officials: Andrius Ališauskas, MD, PhD, Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- Kaunas Hospital of the Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
1) demographic data; 2) medical history (including CHF aetiology, duration, comorbidities, prior hospitalizations, prior procedures, and current pharmacotherapy); 2) physical examination data; 3) anthropometric measurements; 4) questionnaire score data (PHQ-9, HADS, MoCA); 5) ECG data; 6) transthoracic echocardiography data; 7) chest X-ray data; 8) blood test dta (e.g., complete blood count, NT-proBNP, creatinine, urea, electrolytes, inflammatory markers, cardiac troponins); 9) information on in-hospital management, including pharmacological therapy and any procedures; 10) patient outcomes after discharge (will be ascertained through the national Electronic Health Services and Cooperation Infrastructure Information System).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2028-11-20; 2033-11-20
Access Criteria: Any researcher upon reasonable request

REFERENCES:
- [Background] Alisauskas A, Dzikeviciute K, Rimsaite U, Naudziunas A, Razvadauskas H, Zinkiene D, Repecka T, Jucevicius J, Sadauskas S. Prognostic Value of Transthoracic Impedance Cardiography, Amino-Terminal Pro-B-Type Natriuretic Peptide Levels, The Six-Minute Walk Test, and Chest X-Ray in Elderly Patients with Chronic Heart Failure: A Comparative Study in Lithuania. Med Sci Monit. 2024 Sep 27;30:e945647. doi: 10.12659/MSM.945647. PMID 39327721
- [Background] Alisauskas A, Naudziunas A, Sadauskas S, Jankauskiene L, Kalinauskiene E, Vanagaite G. Single-Center Study in Lithuania to Evaluate the Role of Transthoracic Impedance Cardiography in the Diagnosis and Outcome Evaluation of 301 Patients with Chronic Heart Failure Exacerbation. Med Sci Monit. 2022 Dec 24;28:e938389. doi: 10.12659/MSM.938389. PMID 36564931
- [Background] Sadauskas S, Naudziunas A, Unikauskas A, Masanauskiene E, Alisauskas A, Baksyte G, Macas A. Diagnostic and Outcome Prediction Value of Transthoracic Impedance Cardiography in Heart Failure Patients During Heart Failure Flare-Ups. Med Sci Monit. 2018 Sep 18;24:6573-6578. doi: 10.12659/MSM.910754. PMID 30227444
- [Background] Trends in survival after a diagnosis of heart failure in the United Kingdom 2000-2017: population based cohort study. BMJ. 2019 Oct 8;367:l5840. doi: 10.1136/bmj.l5840. No abstract available. PMID 31594775
- [Background] Jones NR, Roalfe AK, Adoki I, Hobbs FDR, Taylor CJ. Survival of patients with chronic heart failure in the community: a systematic review and meta-analysis. Eur J Heart Fail. 2019 Nov;21(11):1306-1325. doi: 10.1002/ejhf.1594. Epub 2019 Sep 16. PMID 31523902
- [Background] Celano CM, Villegas AC, Albanese AM, Gaggin HK, Huffman JC. Depression and Anxiety in Heart Failure: A Review. Harv Rev Psychiatry. 2018 Jul/Aug;26(4):175-184. doi: 10.1097/HRP.0000000000000162. PMID 29975336
- [Background] Li X, Zhou J, Wang M, Yang C, Sun G. Cardiovascular disease and depression: a narrative review. Front Cardiovasc Med. 2023 Nov 21;10:1274595. doi: 10.3389/fcvm.2023.1274595. eCollection 2023. PMID 38084332
- [Background] Reina-Couto M, Pereira-Terra P, Quelhas-Santos J, Silva-Pereira C, Albino-Teixeira A, Sousa T. Inflammation in Human Heart Failure: Major Mediators and Therapeutic Targets. Front Physiol. 2021 Oct 11;12:746494. doi: 10.3389/fphys.2021.746494. eCollection 2021. PMID 34707513
- [Background] Celano CM, Daunis DJ, Lokko HN, Campbell KA, Huffman JC. Anxiety Disorders and Cardiovascular Disease. Curr Psychiatry Rep. 2016 Nov;18(11):101. doi: 10.1007/s11920-016-0739-5. PMID 27671918
- [Background] Moradi M, Doostkami M, Behnamfar N, Rafiemanesh H, Behzadmehr R. Global Prevalence of Depression among Heart Failure Patients: A Systematic Review and Meta-Analysis. Curr Probl Cardiol. 2022 Jun;47(6):100848. doi: 10.1016/j.cpcardiol.2021.100848. Epub 2021 Mar 30. PMID 34006389
- [Background] Chouairi F, Fuery MA, Mullan CW, Caraballo C, Sen S, Maulion C, Wilkinson ST, Surti T, McCullough M, Miller PE, Pacor J, Leifer ES, Felker GM, Velazquez EJ, Fiuzat M, O'Connor CM, Januzzi JL, Desai NR, Ahmad T. The Impact of Depression on Outcomes in Patients With Heart Failure and Reduced Ejection Fraction Treated in the GUIDE-IT Trial. J Card Fail. 2021 Dec;27(12):1359-1366. doi: 10.1016/j.cardfail.2021.06.008. Epub 2021 Jun 22. PMID 34166799
- [Background] Polikandrioti M, Goudevenos J, Michalis LK, Koutelekos J, Kyristi H, Tzialas D, Elisaf M. Factors associated with depression and anxiety of hospitalized patients with heart failure. Hellenic J Cardiol. 2015 Jan-Feb;56(1):26-35. PMID 25701969
- [Background] Di Palo KE. Psychological Disorders in Heart Failure. Cardiol Clin. 2022 May;40(2):269-276. doi: 10.1016/j.ccl.2021.12.014. PMID 35465900
- [Background] Savarese G, Becher PM, Lund LH, Seferovic P, Rosano GMC, Coats AJS. Global burden of heart failure: a comprehensive and updated review of epidemiology. Cardiovasc Res. 2023 Jan 18;118(17):3272-3287. doi: 10.1093/cvr/cvac013. PMID 35150240
- [Background] Rees OL, Wheen P, Anderson LJ. Updates in heart failure. Clin Med (Lond). 2023 Sep;23(5):432-436. doi: 10.7861/clinmed.2023-2023-23.5.Cardio1. PMID 37775162